CLINICAL TRIAL: NCT01679132
Title: BAROSTIM NEO Hypertension Pivotal Trial
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Company resources only allows adequate oversight for one pivotal trial at a time
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360039
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BAROSTIM NEO System (Experimental): Subjects implanted with the BAROSTIM NEO System.
  Interventions: Device: BAROSTIM NEO System and Medical Management

INTERVENTIONS:
Device: BAROSTIM NEO System and Medical Management — Experimental: Device and Medical Management
  Subjects have been implanted with the BAROSTIM NEO System and receive optimal medical management, including drugs to be determined by the subject's physician. Drug types include: Loop Diuretics; Thiazide Diuretics; Potassium-sparing Diuretics; Aldosterone receptor blockers; Beta-blockers; Beta-blockers with intrinsic sympathomimetic activity; Combined alpha- and beta-blockers; ACE inhibitors; Angiotensin II antagonists; Calcium channel blockers- non-Dihydropyridines; Calcium channel blockers- Dihydropyridines; Alpha1-blockers; Central alpha2-agonists and other centrally acting drugs; Direct vasodilators.
  Other Names: Neo System

SUMMARY:
The purpose of this clinical investigation (NCT01679132) is to assess the long-term safety and efficacy of the BAROSTIM NEO System in subjects currently participating in the BAROSTIM Hypertension Pivotal Trial (G120137).

DETAILED DESCRIPTION:
The BAROSTIM NEO Hypertension Trial is a prospective, randomized, controlled trial assessing the safety and efficacy of the BAROSTIM NEO System in subjects with resistant hypertension.

All subjects are now in long term follow-up and are required to have at least one annual visit.

Parameters assessed during visits are:

* Office Cuff Blood Pressure
* Physical Assessment
* Subject Medications
* Serious adverse events

ELIGIBILITY:
Inclusion Criteria:

* Actively participating in the Barostim Hypertension Pivotal Trial and currently implanted with the BAROSTIM NEO device with the device turned ON.
* Have signed a revised approved informed consent form for continued participation in this study.

Exclusion Criteria:

* Treating physician decision that the subject should not continue with therapy.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04-12; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To assess long-term adverse events in subjects implanted with the BAROSTIM NEO System. | For the duration of the study, up to ten years.
  Ascertain the type, frequency, severity and timing of long-term adverse events in G120137 study subjects implanted with the device, while providing a viable treatment option to patients currently implanted with the CVRx BAROSTIM NEO System.

CONTACTS AND LOCATIONS:
Overall Officials: George Bakris, MD, Study Chair — The University of Chicago Medicine; John Bisognano, MD, Study Chair — University of Rochester; Fred Weaver, MD, Study Chair — Keck School of Medicine of the University of Southern California; William Abraham, MD, Study Chair — Ohio State University
Locations (11):
- United States (11):
  - Arizona Heart Rhythm Research Center, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - George Washington University, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Michigan CardioVascular Institute, Saginaw, Michigan
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Aspirus Wausau Hospital, Wausau, Wisconsin